CLINICAL TRIAL: NCT04153240
Title: Positional Therapy for Obstructive Sleep Apnoea: a Randomised Controlled Trial to Assess the Effect on Health and Wellbeing in Older and Younger People
Brief Title: The POSA Trial - Positional Therapy for Positional OSA
Acronym: POSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 252494
Record Dates: First submitted 2019-09-02; First posted 2019-11-06 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Sleep Apnea, Obstructive; Positional Sleep Apnea
Keywords: Positional Therapy; Quality of Life
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective randomised, parallel, double-blinded trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Devices are pre-programmed and by the central site by an unblinded researcher. Devices are allocated randomly by an online randomisation schedule. Researchers and participants, and the central Sleep Therapist remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Positional Therapy (Experimental): The Night Shift™ Sleep Positioner (Advanced Brain Monitoring, USA) - set in 'THERAPY' mode (ie. vibration feedback will be given in response to supine position)
  Interventions: Device: The Night Shift™ Sleep Positioner (Advanced Brain Monitoring, USA)
- Sham Positional Therapy (Sham Comparator): The Night Shift™ Sleep Positioner (Advanced Brain Monitoring, USA) - set in 'MONITOR' mode (ie. no vibration feedback will be given)
  Interventions: Device: The Night Shift™ Sleep Positioner (Advanced Brain Monitoring, USA)

INTERVENTIONS:
Device: The Night Shift™ Sleep Positioner (Advanced Brain Monitoring, USA) — The Night Shift™ Sleep Positioner (Advanced Brain Monitoring, USA) has been developed for adult patients with positional OSA, and snorers. Worn on the back of the neck, it begins to vibrate when the patient starts to sleep in the supine position and increases in intensity until the patient changes.
  Other Names: Positional Therapy

SUMMARY:
Vibro-tactile feedback may be beneficial for some patients, who have positional obstructive sleep apnoea (OSA).

Aim: to determine whether Positional Therapy, applied by a discrete neck-worn vibro-tactile feedback device, is an effective treatment for positional OSA, in reducing the disease severity and associated symptoms, compared to Sham-Positional Therapy. The interaction between treatment and age will also be assessed, since pathophysiology, symptoms and treatment tolerance varies with age.

Methods: A prospective randomised, parallel, double-blinded trial comparing Positional Therapy (Night Shift™; Advanced Brain Monitoring, USA) with Sham-Positional Therapy, performed in older (>65 years) and younger patients with positional OSA (apnoea/hypopnea index (AHI)>5 events/hour, 2:1 when supine). The primary endpoint, AHI at 3 months, will be measured by a repeat study with the device in situ, and compared between Positional Therapy and Sham-Positional Therapy. Patients' subjective symptoms, wellbeing and quality of life, will be assessed by questionnaires at baseline and 3 months. Adherence to therapy will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Ability and willingness to provide informed consent
* AHI >5 events/hour (AASM 2012 scoring criteria) with events occurring at a frequency of 2:1 when supine, compared to non-supine; total % supine sleep >20, <90% of total sleep; central apnoeas <20% total apnoeas; recording of ≥4 hours of analysable signals
* Ability to fit and tolerate wearing the device around the neck during treatment demonstration and initiation

Exclusion Criteria:

* Unstable cardiac disease
* Cardiac arrhythmia corrected with an artificial pacemaker
* Supplemental oxygen
* Secondary sleep pathology e.g. Periodic Limb Movement Syndrome, Narcolepsy, Circadian Disorder, Obesity Hypoventilation Syndrome; or shift workers
* Concerns about sleepy driving or any other potentially dangerous symptom from physician
* BMI ≥40 Kilogram/m2
* Inability to sleep in a non-supine position
* Skin sensitivity or an open wound around neck
* Neck circumference <12inches (30cm) or > 22inches (55cm)
* Tics or tremors of the head
* Sleep with head in upright position
* A female of child-bearing potential that is pregnant or intends to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in OSA severity defined by Apnoea-Hypopnoea Index (AHI): Final AHI after 3 months (adjusted for baseline AHI) of patients treated with Positional Therapy, compared to Sham-Positional Therapy(events/hour) | 3 months
  Apnoea-hypopnea Index (AHI) (events/hour) measured by overnight polygraphy; 0 to <5 events/hour is no OSA, >=5 to <15 events/hour is mild OSA, >=15to <30 events/hour is moderate OSA, >=30 events/hour is severe OSA; Lower AHI is an improvement in disease

SECONDARY OUTCOMES:
Change in AHI (events/hr) in younger (18-<65yrs) compared to older (>=65years) patients: Final AHI after 3 months (adjusted for baseline AHI) of patients treated with Positional Therapy, compared to Sham-Positional Therapy, in older compared to younger | 3 months
  Apnoea-hypopnea Index (AHI) (events/hour) measured by overnight polygraphy; 0 to <5 events/hour is no OSA, >=5 to <15 events/hour is mild OSA, >=15to <30 events/hour is moderate OSA, >=30 events/hour is severe OSA; Lower AHI is an improvement in disease
Changes in Subjective sleepiness: Final scores after 3 months (adjusted for baseline scores) of patients treated with Positional Therapy, compared to sham-treated controls, in Epworth Sleepiness Scale (ESS) | 3 months
  Epworth Sleepiness Scale; 8 scenarios with the likeliness of falling asleep scored in each scenario from 0-3. The 8 Likert response items are summed to calculate a total score. Score range is 0 -24, with higher scores indicating greater daytime sleepiness. Scores >=11 are generally considered abnormal, or positive for excessive daytime sleepiness (EDS).
Changes in Quality of Life - measured by Functional Outcomes of Sleep Questionnaire (FOSQ); Final scores after 3 months (adjusted for baseline scores) of patients treated with Positional Therapy, compared to sham-treated controls, in FOSQ | 3 months
  Functional Outcomes of Sleep Questionnaire (FOSQ) contains 30 items with 5 subscales (scored from 0-4 or 0-6 each). an average score is calculated for each subscale, and the 5 subscales are totaled to produce a total score.Score range is 5-20 points, with higher scores indicating better functional status.
Changes in Anxiety and Depression: Final scores after 3 months (adjusted for baseline scores) of patients treated with Positional Therapy, compared to sham-treated controls, in the Hospital Anxiety and Depression Scale (HADS) | 3 months
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Scores of 8-10 indicate mild disease; 11-14 moderate and 15 to 21 severe. A reduction is considered an improvement in Anxiety or Depression.
Changes in Independent Functioning: Final scores after 3 months (adjusted for baseline scores) of patients treated with Positional Therapy, compared to sham-treated controls, in Townsend Disability Scale | 3 months
  The Townsend disability scale (McGee et al., 1998) is a short index of activities that assesses physical ability in social terms. The scale consists of nine questions or 'items'. The valid responses - 'yes, with no difficulty', 'yes, with some difficulty' and 'no, needs help'-score 0, 1 and 2 respectively. The scale gives equal weighting to each item. Townsend formed groups to interpret the scale (Townsend, 1979): a total score of 0 was regarded as indicating no disability, 1-2 being slightly affected, 3-6 having some disability, 7-10 having appreciable disability, 11-14 having severe disability and 15-18 having very severe disability.
Changes in Quality of Life measured by the Short-form 36 (SF-36); Final scores after 3 months (adjusted for baseline scores) of patients treated with Positional Therapy, compared to sham-treated controls, in SF-36 | 3 months
  The SF-36 questionnaire has 36 items dividing into 8 scales and then again into 2 components (mental and physical). The SF-36 consists of 8 scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Sores out of 100 are presented for the 8 scales and 2 components
Changes in subjective sleep quality and bed partner's perspective: Final scores after 3 months (adjusted for baseline scores) of patients treated with Positional Therapy, compared to sham-treated controls, in Pittsburgh Sleep Quality Index (PSQI) | 3 months
  Pittsburgh Sleep Quality Index (PSQI): 19 items across 7 components are included in scoring. 5 additional items, to be completed by a bed partner, are included in the questionnaire but are not used for scoring. Each of the 7 component scores is determined based on scoring algorithms, with the 7 component scores each yielding a score of 0 -3. A PSQI global (total) score is obtained by summing each of the 7 component scores. Scoring algorithms for each component involve a mixture of averaging Likert response scores, categorization of free text responses (e.g., sleep latency of 15-30 minutes = 1 point), and arithmetic determination of sleep efficiency based on free-text responses. Score range is 0 -21 points, with higher scores indicating better sleep quality.
Changes in Healthcare Utilisation measured by a Healthcare Utilisation Questionnaire | 3 months
  • Final scores after 3 months (adjusted for baseline scores) of patients treated with Positional Therapy, compared to sham-treated controls, in Healthcare Utilisation Questionnaire
Comfort and tolerance of the Positional Therapy device | 3 months
  • Visual analogue scale (VAS) of comfort and tolerance of device. The scale is a 100mm line with 0 representing low comfort and tolerance and 100 representing high comfort and tolerance
Adherence to Positional Therapy measured by the Night Shift device | 3 months
  • Adherence to positional therapy measured by the Night Shift device will be reported as mean hrs/night over the entire 3 months. Good adherence for other OSA therapies, including CPAP, is suggested by an arbitrary threshold over >4 hours/night.
Changes to Sleeping position measured by the Night Shift device on the first (monitoring night) and last night of Therapy | 3 months
  • A change from baseline to 3 months post Positional Therapy, compared to sham-treated controls NightShift data:
  - percentage supine sleep compared to total sleep time (in previous populations, a reduction of supine sleep time by 84% is a good outcome)
  A reduction in the supine sleep is an improvement
Changes in sleep-disordered breathing measured by overnight polygraphy | 3 months
  • A change from baseline to 3 months post Positional Therapy, compared to sham-treated controls, in oxygenation measured by:
  -oxygen desaturation index (ODI; events/hour); measured by the number of overnight desaturations >3% and >4% as an index per hour An improvement is indicated by a reduction in ODI (normal is <5 events/hr)

OTHER OUTCOMES:
Effect of age on treatment effect, and on changes in AHI | 3 months
  A change from baseline to 3 months post Positional Therapy, compared to sham-treated controls, in older compared to younger patients in AHI

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Churchill Hospital, Oxford, Oxfordshire
  - Aintree Hospital, Liverpool
  - The Royal Free Hospital, London
  - Royal Brompton Hospital, London
  - The Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kelly JL, Turnbull CD, Newson R, Dobson M, Hedley EL, ALQarni AS, Nevinson A, Dawson D, Nickol A, West S, Talbot NP, Rahman NM, Stradling J, Morrell MJ; POSA trial investigators. Vibrotactile positional therapy for the treatment of positional obstructive sleep apnoea: a multicentre, randomised controlled trial. Thorax. 2025 Sep 24:thorax-2024-222681. doi: 10.1136/thorax-2024-222681. Online ahead of print. PMID 40992934